CLINICAL TRIAL: NCT01067014
Title: The iO-Flex® Study: Evaluation of the Baxano iO-Flex® System for Decompressive Lumbar Surgery
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Baxano Surgical, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CP-1318
Record Dates: First submitted 2010-02-09; First posted 2010-02-11 (Estimated); Last update posted 2013-09-23 (Estimated); Status verified 2013-09

CONDITIONS: Lumbar Spinal Stenosis
Keywords: Lumbar spinal stenosis; Decompression; Lumbar spinal decompression; Lumbar spinal decompressive surgery
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- iO-Flex
  Interventions: Device: Baxano iO-Flex® System

INTERVENTIONS:
Device: Baxano iO-Flex® System — Decompressive lumbar surgery using Baxano iO-Flex® System

SUMMARY:
The purpose of this study is to evaluate the clinical performance of the iO-Flex® System in reducing pain and symptom severity in patients with one or two level lumbar spinal stenosis that requires surgery.

ELIGIBILITY:
Inclusion Criteria

Candidates for this study must meet ALL of the following criteria:

1. Age ≥18 years
2. Leg/buttock pain with or without back pain
3. Failed nonoperative medical management
4. A minimum leg pain score of 4.0 cm on the Visual Analogue Scale (VAS)
5. Clinical/radiographic diagnosis of LSS in the L2-L3 to L5-S1 region
6. Able and willing to give voluntary, written informed consent to participate in this clinical study

Exclusion Criteria

Candidates will be excluded from the evaluation if ANY of the following apply:

1. Back pain only
2. A diagnosis of central stenosis only
3. More than two levels requiring decompression
4. Fixed motor deficit
5. Significant instability of the lumbar spine as defined by ≥ 4mm translation between standing flexion and extension lumbar spine plain film radiographs
6. Sustained pathologic fractures of the vertebrae or multiple fractures of the vertebrae and/or hips
7. Primary disc pathology and/or patients who will undergo a discectomy
8. Prior surgery of the lumbar spine at the level(s) of planned treatment
9. Spondylolisthesis or degenerative spondylolisthesis greater than Grade 1 (on a scale of 1 to 4)
10. Spondylolysis (pars fracture) at any level in the lumbar spine
11. Degenerative lumbar scoliosis with a Cobb angle greater than or equal to 25°
12. Symptomatic vascular claudication in the lower extremities
13. Cauda equina syndrome (neural compression causing neurogenic bowel or bladder dysfunction)
14. Evidence of active (systemic or local) infection at time of surgery
15. Paget's disease at involved segment or metastasis to the vertebra, osteomalacia, or other metabolic bone disease
16. Tumor in the spine or a malignant tumor except for basal cell carcinoma
17. Prisoner or transient
18. Recent history of known narcotic abuse
19. Any significant psychological disturbance past or present, psychotic or neurotic, that could impair the consent process or ability to complete subject self-report questionnaires
20. Involved in pending litigation of the spine or worker's compensation related to the back
21. Inability to communicate clearly in the English language
22. Morbid obesity (BMI > 40)
23. Plans to relocate within the next 2 years
24. Pregnant or planning to become pregnant
25. Irreversible coagulopathy or bleeding disorder

    a. Subjects on Coumadin or other anticoagulants may participate. Investigators should follow routine practices for perioperative discontinuation and reinitiation of anticoagulants.
26. Subject unwilling to undergo blood transfusion, if necessary

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at least 18 years of age presenting with failed conservative treatment for one or two level lumbar spinal stenosis
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2010-02; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Change in the Symptom Severity domain of the Zurich Claudication Questionnaire (ZCQ) from baseline to 6 months post-procedure quantified as a percentage of subjects with an improvement of at least 0.5 points | 6 months
Change in Visual Analog Scale (VAS) for leg pain related to lumbar spinal stenosis at the treatment level from baseline to 6 months post-procedure quantified as a percentage of subjects with an improvement of at least 30% | 6 months
Re-operation at the treatment level(s) at one year post-procedure | One year
Acute safety outcomes will be determined by evaluating the type, frequency, severity, and relatedness of adverse events through discharge visits for all subjects | Hospital discharge

SECONDARY OUTCOMES:
Changes in Visual Analog Scale scores compared to baseline | 6 weeks, 3 months, 6 months, 12 months, 24 months
Changes in Zurich Claudication Questionnaire scores compared to baseline | 6 weeks, 3, 6, 12, and 24 months
Changes in Oswestry Disability Index scores compared to baseline | 6 weeks, 3, 6, 12, and 24 months
Flexion/extension lumbar spine plain film radiographs will be collected and assessed for presence/absence of instability at baseline, 6-month, 12-month, and 24-months | 6, 12, and 24 months
Long term safety outcomes that occur after discharge through 2 years post-procedure will be determined by evaluating adverse events involving the musculoskeletal or neurological systems | Through 2 years

CONTACTS AND LOCATIONS:
Locations (18):
- United States (18):
  - Eden Medical Center, Castro Valley, California
  - Olympia Medical Center, Los Angeles, California
  - Watsonville Community Hospital, Watsonville, California
  - Resurgens Orthopaedics, Cumming, Georgia
  - Suburban Orthopedics, Bartlett, Illinois
  - Spine Midwest, Inc., Jefferson City, Missouri
  - McCune-Brooks Regional Hospital, Joplin, Missouri
  - Buffalo Spine Surgery, Lockport, New York
  - Triangle Orthopaedic Associates, Chapel Hill, North Carolina
  - Moses Cone Hospital, Greensboro, North Carolina
  - Caldwell Memorial Hospital, Lenoir, North Carolina
  - Rothman Institute, Bensalem, Pennsylvania
  - Easton Hospital, Easton, Pennsylvania
  - Carolina Neurosurgery & Spine Center, Greenwood, South Carolina
  - Neurospine Solutions, PC, Bristol, Tennessee
  - Spine Works Institute, North Richland Hills, Texas
  - University of Utah, Salt Lake City, Utah
  - Tuckahoe Orthopaedic Associates, Richmond, Virginia